CLINICAL TRIAL: NCT01220232
Title: Open-Label, Fixed-Sequence, Crossover Study To Estimate The Effect Of Lersivirine On The Pharmacokinetics Of Abacavir/Lamivudine In Healthy Subjects
Brief Title: Estimate The Effect Of Lersivirine On The Pharmacokinetics Of Abacavir/Lamivudine In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5271048
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Volunteers
Keywords: Lersivirine; UK-453; 061; NNRTI; Abacavir; Lamivudine; Combivir; Pharmacokinetics; Drug Interaction; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — abacavir, lamivudine drug combination; UK 453,061

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abacavir/Lamivudine (Active Comparator)
  Interventions: Drug: Abacavir/Lamivudine
- Lersivirine + Abacavir/Lamivudine (Experimental)
  Interventions: Drug: Abacavir/Lamivudine; Drug: Lersivirine

INTERVENTIONS:
Drug: Abacavir/Lamivudine — Abacavir/Lamivudine 600/300 mg QD for 5 days
  Arms: Abacavir/Lamivudine
Drug: Abacavir/Lamivudine — Abacavir/Lamivudine 600/300 mg QD for 10 days
  Arms: Lersivirine + Abacavir/Lamivudine
Drug: Lersivirine — Lersivirine 750 mg QD for 10 days
  Arms: Lersivirine + Abacavir/Lamivudine

SUMMARY:
This will be an open-label, fixed-sequence, multiple dose crossover study in 14 healthy male and/or female subjects, to estimate the effect of steady state lersivirine on the steady state pharmacokinetics of abacavir/lamivudine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* History of hypersensitivity to abacavir, lamivudine and/or lersivirine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To estimate the effect of steady state lersivirine 750 mg on the steady state pharmacokinetics of abacavir/lamivudine. | 17 days

SECONDARY OUTCOMES:
To investigate the safety and tolerability of lersivirine when co-administered with abacavir/lamivudine. | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271048&StudyName=Estimate%20The%20Effect%20Of%20Lersivirine%20On%20The%20Pharmacokinetics%20Of%20Abacavir/Lamivudine%20In%20Healthy%20Subjects%20